CLINICAL TRIAL: NCT02141581
Title: Vaccination and Infection: Indicators of Immunological Health and Responsiveness. Project 1: Plasmablast Trafficking and Antibody Response in Influenza Vaccination;
Brief Title: Plasmablast Trafficking and Antibody Response in Influenza Vaccination (SLVP021 2011-2014)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Professor, Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SU-21987- 2011; 1U19AI090019-01 (NIH)
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Influenza
Keywords: Intramuscular inactivated trivalent influenza vaccine; Intradermal inactivated trivalent influenza vaccine; Live, attenuated influenza vaccine; Young adults
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A Fluzone® (IM) (Experimental): Participants in this group will be randomized to the trivalent inactivated influenza vaccine (TIV), Fluzone®, administered intramuscularly (IM)
  2011-2012, 2012-2013 or 2013-2014 Fluzone was used as appropriate for the current year of study
  Interventions: Biological: Fluzone® (IM)
- Group B Fluzone® Intradermal (ID) (Experimental): Participants in this group will be randomized to the trivalent inactivated influenza vaccine (TIV), Fluzone® Intradermal, administered intradermally (ID)
  2011-2012, 2012-2013 or 2013-2014 Fluzone Intradermal was used as appropriate for the current year of study
  Interventions: Biological: Fluzone® Intradermal (ID)
- Group C 2011-2012 FluMist® (Experimental): Participants in this group will be randomized to 2011-2012 live attenuated influenza vaccine, FluMist®, administered intranasally.
  FluMist was only used in the first year of study.
  Interventions: Biological: 2011-2012 FluMist®

INTERVENTIONS:
Biological: Fluzone® (IM) — This vaccine is given intramuscularly (IM)
  Other Names: Trivalent inactivated influenza vaccine (TIV); FDA-licensed seasonal influenza vaccine
  Arms: Group A Fluzone® (IM)
Biological: Fluzone® Intradermal (ID) — This vaccine is given intradermally (ID)
  Other Names: Trivalent inactivated influenza vaccine (TIV); FDA-licensed seasonal Influenza Vaccine
  Arms: Group B Fluzone® Intradermal (ID)
Biological: 2011-2012 FluMist® — This vaccine is given intranasally
  Other Names: Live, attenuated influenza vaccine (LAIV); FDA-licensed seasonal influenza vaccine
  Arms: Group C 2011-2012 FluMist®

SUMMARY:
The purpose of this study is to investigate the responses to licensed trivalent, inactivated influenza vaccine (TIV) delivered by different routes: intramuscular (IM) and intradermal (ID) and to the live, attenuated influenza vaccine (LAIV) administered intranasally -- all given to generally healthy male and female adult volunteers.

DETAILED DESCRIPTION:
The aim of this study is to compare the response to different formulations of licensed influenza vaccines.

The type of seasonal influenza vaccination(s) received independently by volunteers in the year(s) since their last study visit will not impact eligibility. Volunteers will be assigned into one of three vaccine groups (intramuscular trivalent inactivated influenza vaccine (TIV); live attenuated influenza vaccine (LAIV- given year 1 only) or intradermal TIV, based on the type of study vaccine they received in 2010, 2011, 2012, or 2013. All participants will receive a single dose of their assigned seasonal influenza vaccine. Volunteers will complete 3 study visits at Day 0, Day 6-8 and Day 24-32.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy, ambulatory between the ages of 8-33 years, inclusively.
* Willing to complete the informed consent process
* Availability for follow-up for the planned duration of the study at least 28 days after immunization
* Acceptable medical history and vital signs

Exclusion Criteria:

* Prior vaccination with seasonal TIV or LAIV
* Prior off-study vaccination with TIV or LAIV in the current flu season
* Allergy to egg or egg products, or to vaccine components or thimerosal (TIV multidose vials only)
* Life-threatening reactions to previous influenza vaccinations
* Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
* Asthma or history of wheezing (for volunteers receiving LAIV only)
* Participants in close contact with anyone who has a severely weakened immune system should not receive LAIV (for volunteers receiving LAIV only)
* History of immunodeficiency (including HIV infection)
* Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease, or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol
* Blood pressure >150 systolic or >95 diastolic at first study visit
* Chronic Hepatitis B or C
* Recent or current use of immunosuppressive medication, including systemic glucocorticoids (corticosteroid nasal sprays, inhaled steroids and topical steroids are permissible in both groups)
* Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia)
* Autoimmune disease (including rheumatoid arthritis) treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol
* History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
* Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except up to 325 mg. aspirin per day), Plavix, or Aggrenox must be reviewed by investigator to determine if this would affect the volunteer's safety
* Receipt of blood or blood products within the past 6 months or planned receipt of blood products prior to completion of study visits
* Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
* Inactivated vaccine 14 days prior to vaccination or planned non-study vaccination prior to completion of Visit 03 (~Day 28 after the study vaccination)
* Live, attenuated vaccine within 60 days of vaccination or planned non-study vaccination prior to completion of Visit 03 (~Day 28 after the study vaccination)
* Need an allergy immunization (that cannot be postponed) during the study period V01 to V03 (~Day 28)
* History of Guillain-Barré Syndrome
* Pregnant or lactating woman
* Use of investigational agents within 30 days prior to enrollment or planned use of investigational agents prior to completion of study visits
* Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment or planned blood donation prior to completion of study visits
* Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol

Ages: 8 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2011-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia L Dekker, MD, Principal Investigator — Stanford University; Harry B Greenberg, MD, Principal Investigator — Stanford University; Xiaosong He, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford LPCH Vaccine Program, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The NIH Human Immunology Project Consortium (HIPC) data repositories (ImmPORT) may store the results of the research assays results. Genetic data that is developed in this study may be made available to other researchers through the National Center for Biotechnology Information (NCBI) databases. Results from research assays will be labeled with a unique ID code and the volunteer identity (except for age) will not be disclosed.

REFERENCES:
- [Background] Vollmers C, Sit RV, Weinstein JA, Dekker CL, Quake SR. Genetic measurement of memory B-cell recall using antibody repertoire sequencing. Proc Natl Acad Sci U S A. 2013 Aug 13;110(33):13463-8. doi: 10.1073/pnas.1312146110. Epub 2013 Jul 29. PMID 23898164
- [Background] He XS, Holmes TH, Sanyal M, Albrecht RA, Garcia-Sastre A, Dekker CL, Davis MM, Greenberg HB. Distinct patterns of B-cell activation and priming by natural influenza virus infection versus inactivated influenza vaccination. J Infect Dis. 2015 Apr 1;211(7):1051-9. doi: 10.1093/infdis/jiu580. Epub 2014 Oct 21. PMID 25336731
- [Background] Le Gars M, Kay AW, Bayless NL, Aziz N, Dekker CL, Swan GE, Davis MM, Blish CA. Increased Proinflammatory Responses of Monocytes and Plasmacytoid Dendritic Cells to Influenza A Virus Infection During Pregnancy. J Infect Dis. 2016 Dec 1;214(11):1666-1671. doi: 10.1093/infdis/jiw448. Epub 2016 Sep 21. PMID 27655870

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A Fluzone® (IM): Participants in this group will be randomized to Fluzone® administered intramuscularly (IM)
- Group B Fluzone® (ID): Participants in this group will be randomized to Fluzone® administered intradermally (ID)
- Group C FluMist®: Participants in this group will be randomized to FluMist® administered intranasally.
Period: Overall Study
Arm/Group | Group A Fluzone® (IM) | Group B Fluzone® (ID) | Group C FluMist®
Started | 42 | 19 | 25
Completed | 42 | 19 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A Fluzone® (IM) | Group B Fluzone® (ID) | Group C FluMist® | Total
Number analyzed (Participants) | 42 | 19 | 25 | 86
Age, Customized [Count of Participants; unit: Participants]
  Age 18-30 years | 32 | 19 | 25 | 76
  Age 8-17 years | 10 | 0 | 0 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 9 | 15 | 49
  Male | 17 | 10 | 10 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 1 | 7
  Not Hispanic or Latino | 39 | 16 | 24 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 10 | 6 | 9 | 25
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 3
  Black or African American | 0 | 0 | 0 | 0
  White | 25 | 10 | 9 | 44
  More than one race | 2 | 1 | 6 | 9
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 19 | 25 | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants From Each Arm Who Received Influenza Vaccine
Time Frame: Baseline to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Group A Fluzone® (IM) | Group B Fluzone® (ID) | Group C Flumist®
Number analyzed (Participants) | 42 | 19 | 25
Participants | 42 | 19 | 25

2. Secondary Outcome: Number of Participants With Related Adverse Events
Description: Number of participants with Related Adverse Events with a 0% Frequency Threshold
Time Frame: Baseline to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Group A Fluzone® (IM) | Group B Fluzone® (ID) | Group C Flumist®
Number analyzed (Participants) | 42 | 19 | 25
Participants
  Bronchospasm | 1 | 0 | 0
  Erythema at injection site | 1 | 0 | 0
  No Related Adverse Events | 40 | 19 | 25

3. Other Pre Specified Outcome: Frequency of Vaccine-specific Antibody Secreting Cells on Day 5 and Day 7 After Vaccination
Time Frame: Baseline to Day 7
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Group A Fluzone® (IM) | Group B Fluzone® (ID) | Group C FluMist®
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/19 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/19 | 1/25
Other Adverse Events (participants affected / at risk) | 3/42 | 3/19 | 2/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A Fluzone® (IM) (N=42) | Group B Fluzone® (ID) (N=19) | Group C FluMist® (N=25)
Panic Attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — Panic attack associated with Bipolar disorder resulting in prolonged hospitalization. Episode not related to vaccination or participation in study.
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Depression leading to hospitalization, not associated with vaccine injection or study participation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A Fluzone® (IM) (N=42) | Group B Fluzone® (ID) (N=19) | Group C FluMist® (N=25)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Associated with vaccine injection. Chest tightness and cough after injection, relieved by inhaler, without sequelae.
Erythema at injection site (General disorders) | 0 (0) | 1 (1) | 0 (0) — Associated with vaccine injection. Erythema resolved without sequelae.
Presyncope (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) — Not associated with vaccine injection. Associated with blood draw. All subjects recovered within 10 minutes of blood draw without sequelae.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No